CLINICAL TRIAL: NCT07151430
Title: Development and Validation of a Comprehensive Management Service Package for Older Adults With Multimorbidity: A Randomized Controlled Trial
Brief Title: Development and Validation of a Comprehensive Management Service Package for Older Adults With Multimorbidity
Acronym: COMPASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, yinchunlin, Director of Department of Cardiology, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XWH-MULTICOMORB-2024-001; 2023YFC3605003 (Other: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Multimorbidity; Hypertension; Diabetes Mellitus; Coronary Artery Disease; Dyslipidemia; Stroke; Arthritis; Cognitive Impairment; Depression - Major Depressive Disorder; Chronic Kidney Disease; Chronic Liver Diseases
Keywords: management service package; multimorbidity; quality of life; intrinsic capacity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Coronary Artery Disease; Dyslipidemias; Stroke; Arthritis; Cognitive Dysfunction; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Comprehensive multimorbidity management service package (digital tools, MDT decision support, lifestyle interventions, long-term management tools).
  Interventions: Device: Service Package Group
- Control Arm (No Intervention): Standard of care without the service package.

INTERVENTIONS:
Device: Service Package Group — patients receive comprehensive multimorbidity management service package (digital tools, MDT decision support, lifestyle interventions, long-term management tools).
  Arms: Experimental Arm

SUMMARY:
This study aims to test a new comprehensive management service package for older adults with two or more chronic conditions (multimorbidity). The package includes digital health tools, personalized guidance, and long-term management support. Researchers will compare the service package with usual care to see whether it reduces hospital readmissions, improves quality of life, and supports daily functioning. About 394 participants will be randomly assigned to either the service package group or the usual care group. Participants will be followed for 6 months to measure health outcomes, treatment adherence, and safety.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if a new comprehensive management service package can help improve health outcomes for older adults who have two or more chronic conditions (multimorbidity). It will also learn about the safety, acceptability, and cost-effectiveness of the service package.

The main questions it aims to answer are:

1. Does the service package lower the number of hospital readmissions in older adults with multimorbidity?
2. Does it improve quality of life, daily function (intrinsic capacity), and treatment adherence?
3. What are the costs and potential risks of using the service package compared to usual care? Researchers will compare the service package to usual care (no service package).

Participants will:

1. Be randomly assigned to either the service package group or the usual care group
2. Use the digital tools and health management support included in the service package (such as apps, monitoring devices, and personalized health guidance)
3. Receive regular follow-up visits and surveys over 6 months to track their health, hospital use, and satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years
2. Diagnosed with ≥2 chronic diseases or geriatric syndromes (e.g., hypertension, diabetes, frailty, depression)
3. Willing to provide informed consent

Exclusion Criteria:

1. Life expectancy <1 year due to severe illness (e.g., cardiogenic shock)
2. Currently participating in other clinical trials

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital readmission rate | 6 months
  Hospital readmission rate

IPD SHARING:
Plan to Share IPD: No